CLINICAL TRIAL: NCT07013591
Title: Randomized Clinical Trial of β Nicotinamide Mononucleotide in Patients Undergoing CABG Surgery
Brief Title: Nicotinamide Mmononucleotide in Patients Undergoing CABG Surgery
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Shalendar Bhasin, MD, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025P000420; 1U01AG089040-01 (NIH)
Record Dates: First submitted 2025-05-09; First posted 2025-06-10 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Coronary Artery Bypass Graft
Keywords: coronary artery bypass graft; cardiac surgery; cardiopulmonary bypass; nicotinamide; NMN; acute kidney injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- NMN (MIB-626) for 7 days preoperatively, on day of surgery, and for 4 days postoperatively (Experimental): NMN (MIB-626) 1000 mg PO daily, for 7 days preoperatively, on day of surgery, and for 4 days postoperatively
  Interventions: Drug: MIB-626
- NMN administered for 2 days preoperatively, on the day of surgery, and for 4 days postoperatively (Experimental): NMN (MIB-626) 1,000 mg PO twice daily, administered for 2 days preoperatively, on the day of surgery, and for 4 days postoperatively
  Interventions: Drug: MIB-626
- Placebo (Placebo Comparator): Placebo administered for 7 days preoperatively, on the day of surgery, and for 4 days postoperatively
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: MIB-626 — An orally-administered stable crystalline tablet formulation of NMN
  Arms: NMN (MIB-626) for 7 days preoperatively, on day of surgery, and for 4 days postoperatively; NMN administered for 2 days preoperatively, on the day of surgery, and for 4 days postoperatively
Other: Placebo — matching placebo tablets
  Arms: Placebo

SUMMARY:
The investigators will perform a phase 2a, randomized, double-blind, placebo-controlled clinical trial in adult patients undergoing elective coronary artery bypass grafting (CABG) surgery to investigate the effects of oral nicotinamide mononucleotide (NMN) administration on myocardial NAD+ concentrations and on postoperative markers of myocardial and kidney injury.

DETAILED DESCRIPTION:
This is a phase 2a, randomized, double-blind, parallel-group, placebo-controlled clinical trial in adult patients undergoing elective coronary artery bypass grafting (CABG) surgery. A total of 90 patients will be randomized 1:1:1 to placebo or to one of two dosing regimens of NMN seven days prior to surgery as follows:

Arm A: NMN 1,000 mg PO twice daily, administered for 7 days preoperatively, on the day of surgery, and for 4 days postoperatively

Arm B: NMN 1,000 mg PO twice daily, administered for 2 days preoperatively, on the day of surgery, and for 4 days postoperatively

Arm C: Placebo PO twice daily, administered for 7 days preoperatively, on the day of surgery, and for 4 days postoperatively

There are two major study aims:

Aim 1: Test the effect of oral NMN administration on myocardial NAD+ concentration.

Aim 2: Test the effect of oral NMN administration on postoperative myocardial and kidney injury parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Scheduled to undergo elective isolated CABG surgery with cardiopulmonary bypass (CPB)
3. At increased risk of postoperative complications based on ≥1 of the following:

   1. Age ≥65 years
   2. eGFR <45 ml/min/1.73m2
   3. Documented history of congestive heart failure or left ventricular ejection fraction (LVEF) ≤40% within 6 months before surgery
   4. Diabetes mellitus and urine albumin-to-creatinine ratio >30 mg/g creatinine
   5. Peripheral arterial disease
   6. Anemia, defined as hemoglobin <10 g/dl
   7. Prior cardiac surgery

Exclusion Criteria:

1. Any of the following laboratory abnormalities at the time of screening:

   1. ALT >3-fold the upper limit of normal
   2. eGFR <30 ml/min/1.73m2 or ESKD on dialysis
   3. Hemoglobin <8 g/dl
2. History of gastric bypass or malabsorption
3. Active alcohol or illicit substance use in the prior 6 months
4. Participation in an investigational trial to evaluate pharmaceuticals or biologics within the past 3 months or 5 half-lives, whichever is shorter
5. Pregnant or breast-feeding
6. Unwillingness to use contraception while taking study drug and for 8 weeks after the last dose for women of reproductive age or non-sterilized male participants who are sexually active with a female partner of childbearing potential
7. Current use of niacin >100 mg/day or NMN, nicotinamide, or nicotinamide riboside at any dose
8. Conflict with other research studies
9. Any condition which, in the judgement of the investigator, might increase the risk to the participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2028-10-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
NAD+ concentration in the myocardial tissue | Intraoperatively (single time point)
  NAD+ concentration in the myocardial tissue (right atrial appendage) obtained intraoperatively, measured using the validated NADome Quant assay

SECONDARY OUTCOMES:
Intracellular levels of NAD+ and related metabolites | Intraoperatively (single time point)
  NAD+, NADH, and related metabolite concentrations in discarded tissue collected intraoperatively, including right atrial appendage, internal mammary artery, sternal muscle, and fat
Circulating levels of NAD+ and related metabolites | Baseline to day 90
  NAD+, NADH, and related metabolite concentrations in the circulation and in peripheral blood mononuclear cells
Markers of cardiac injury/dysfunction | Preoperatively, on ICU arrival, and on postoperative days 1-4
  Circulating levels of cardiac troponin I, creatine kinase MB fraction (CKMB), and N-terminal pro-B-type natriuretic peptide (NT-pro-BNP)
Acute kidney injury (AKI) | 7 days post-operatively
  Incidence of acute kidney injury (AKI) defined according to the Kidney Disease Improving Global Outcomes (KDIGO) criteria as any of the following: 1) urine output <0.5 ml/kg/h for ≥6 consecutive hours (assessed within the first 48h or until the Foley catheter is removed, whichever occurs first); 2) an increase in SCr ≥0.3 mg/dl within the first 48h; 3) an increase in SCr ≥50% within the first 7 days; or 4) receipt of KRT within the first 7 days
Serum creatinine (SCr) | Immediately pre-operative to 7 days post-operative
  Maximum baseline-adjusted changes in SCr
Cystatin C | Preoperatively, on ICU arrival, and on postoperative days 1-4
  Circulating levels of cystatin C
Neutrophil gelatinase-associated lipocalin (NGAL) | Preoperatively, on ICU arrival, and on postoperative days 1-4
  Circulating levels of measured neutrophil gelatinase-associated lipocalin (NGAL)
Kidney Injury Molecule-1 (KIM-1) | Preoperatively, on ICU arrival, and on postoperative days 1-4
  Circulating levels of KIM-1
NMN level | Preoperatively, on ICU arrival, and on postoperative days 1-4
  Plasma concentrations of NMN
2PY Level | Preoperatively, on ICU arrival, and on postoperative days 1-4
  Plasma concentrations of 2PY
N-Methylnicotinamide level | Preoperatively, on ICU arrival, and on postoperative days 1-4
  Plasma N-methylynicotinamide level
nicotinamide level | Preoperatively, on ICU arrival, and on postoperative days 1-4
  Plasma nicotinamide concentrations

OTHER OUTCOMES:
Left ventricular ejection fraction (LVEF) | change from immediately preoperative to immediate postoperative
  Left ventricular ejection fraction (LVEF) measured by a transesophageal echocardiogram (TEE)
Atrial fibrillation | First seven days postoperatively
  Frequency of new-onset atrial fibrillation. Atrial fibrillation must be confirmed on a 12-lead ECG or a rhythm strip, confirmed by a healthcare provider, or treated (either medically [e.g., amiodarone] or with electrical cardioversion)
Vasoactive-inotropic score | Immediately preoperatively to 24-hours post-incision
  The vasoactive-inotropic score is a validated method for integrating all vasoactive medications and their doses on an hourly basis into a single measure. The score ranges from 0 to 100, with higher scores indicating greater cardiovascular support needs.
Time-to-liberation from vasoactive medications | End of cardiopulmonary bypass to 24 hours post surgery
  Time (in hours) from end of cardiopulmonary bypass (CPB) to liberation from all vasopressors and inotropes.
ICU length of stay | Time in days in the ICU post-operatively, from the day of admission to the ICU postoperatively after the coronary artery bypass surgery to the time of release from ICU or date of death from any cause, up to 90 days
  time to release from the ICU post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Shalender Bhasin, MB, BS, Principal Investigator — Brigham and Women's Hosptial
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with the NIH Policy for Data Management and Sharing, as well as the NIH Genomic Data Sharing Policy, deidentified data generated from this research will be shared with the research community by depositing it in the Harvard Dataverse. This will include any large-scale genomic data generated.
Supporting Information: Study Protocol, ICF
Time Frame: Within 1 year of the end date of the study
Access Criteria: Only de-identified data will be available for scientific research upon review of specific request and provision of IRB-approval.